CLINICAL TRIAL: NCT03241914
Title: Megestrol Acetate Plus LNG-IUS to Megestrol Acetate in Young Women With Early Endometrial Cancer
Brief Title: Megestrol Acetate Plus LNG-IUS in Young Women With Early Endometrial Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Principal Investigator, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-30-2
Record Dates: First submitted 2017-07-12; First posted 2017-08-08 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Endometrial Neoplasm Malignant Stage I
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Megestrol Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MA (Active Comparator): Patients will receive megestrol acetate 160 mg by mouth daily for at least 3 months.Then every 3 months, an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Drug: Megestrol Acetate
- MA+LNG-IUS (Experimental): Patients will receive MA (160mg po qd) plus LNG- IUS insertion for at least 3 months. Then every 3 months, an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Drug: Megestrol Acetate; Device: Levonorgestrel-releasing Intrauterine System(LNG-IUS)

INTERVENTIONS:
Drug: Megestrol Acetate — At a dosage of 160 mg/day
  Other Names: Megace
Device: Levonorgestrel-releasing Intrauterine System(LNG-IUS) — levonorgestrel 52mg. It is a hormone-releasing T-shaped intrauterine system.
  Other Names: Mirena Intrauterine Device; Mirena
  Arms: MA+LNG-IUS

SUMMARY:
To see if megestrol acetate plus Levonorgestrel-releasing intrauterine system (LNG-IUS) will not be inferior to returning the endometrial tissue to a normal state than megestrol acetate alone in patients with early endometrial cancer.

DETAILED DESCRIPTION:
After diagnosed of endometrioid endometrial cancer (EEC) by hysteroscopy, patients will be enrolled. Age, waist circumstances, blood pressure, basic history of infertility, blood pressure, serum lipid level and side effects will be collected. Blood tests, including fasting blood glucose (FBG), postprandial blood glucose (PBG), fasting insulin (FINS), SHBG, sex hormone levels, blood lipids and anti-müllerian hormone(AMH) will be performed before treatment to evacuate their metabolic conditions.

Patients are randomized to 1 of 2 treatment groups. Patients will receive MA (megestrol acetate) 160 mg by mouth daily for at least 3 months on Arm I. Patients will receive MA 160 mg plus LNG-IUS insertion for at least 3 months on Arm II. Then an hysteroscope will be used to evaluate the endometrial condition every 3 months, and the findings will be recorded. For patients with EEC, complete response (CR) is defined as the reversion of endometrial disease to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia without atypic or atypical hyperplasia; no response (NR) is defined as the persistence of the disease; and progressive disease (PD) is defined as the progression of endometrial lesions. Continuous therapies will be needed in PR, NR or PD.

As the reason of the low response rate of LNG-IUS alone in EC patients (nearly 50%), and the potential limitation of LNG-IUS to focal cancer lesion in endometrial cavity, the investigators did not add LNG-IUS alone as a single control group.

After completion of study treatment, 2 months of maintenance treatment will be recommended for patients with CR, and participants will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Primarily have a confirmed diagnosis of endometrioid endometrial cancer based upon hysteroscopy
* MRI parameters shows there's no myometrial invasion, extension beyond corpus, or enlarged lymph nodes
* Have a desire for remaining reproductive function or uterus
* Need to be able to undergo correlative treatment and follow-up

Exclusion Criteria:

* Acute liver disease or liver tumor (benign or malignant) or renal dysfunction
* Pregnancy or suspicion of pregnancy
* Have a history of EAH or EC and have disease relapse during Merina insertion
* Under treatment of high-dose progestin therapy more than 3 months in recent 6 months
* Congenital or acquired uterine anomaly including fibroids if they distort the uterine cavity
* Confirmed diagnosis of malignant tumor in genital system
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* Hypersensitivity or contradiction to any component of this product
* Ask for removal of the uterus or other conservative treatment
* Smoker(>15 cigarettes a day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Pathological response rate | From date of randomization until the date of CR or date of hysterectomy, whichever came first, assessed up to 12 months
Pathological response time | From date of randomization until the date of CR or date of hysterectomy, whichever came first, assessed up to 12 months
  median time of histologic regression from endometrial atypical hyperplasia to benign endometrium

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 2 years after the treatment for each patient
  Common side effects from these drugs include weight gain, vaginal spotting and descent of sexuality. Severe side effects include thrombus and diseases related. The investigators will record any mental or body symptoms and evaluate the correlation.
Rate of relapse | up to 2 years after the treatment for each patient
Rate of pregnancy | up to 2 years after the treatment for each patient
Compliance | up to 2 years after the treatment for each patient
  The investigators designed a questionnaire to evaluate the compliance through treatment as side effects of oral megestrol acetate may be more common than LNG-IUS. Self Efficacy, physical activity and social support will be scored (1 to 5) and compared between different arms.

OTHER OUTCOMES:
Economic consequences through study completion | From date of randomization until the date of CR or date of hysterectomy, whichever came first, assessed up to 12 months
  The investigators will evaluate whether the combination could shorten therapeutic period, so that bring economic benefits to the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu Z, Yang B, Guan J, Shan W, Liao J, Shao W, Chen X. Comparison of the effect of oral megestrol acetate with or without levonorgestrel-intrauterine system on fertility-preserving treatment in patients with early-stage endometrial cancer: a prospective, open-label, randomized controlled phase II trial (ClinicalTrials.gov NCT03241914). J Gynecol Oncol. 2023 Jan;34(1):e32. doi: 10.3802/jgo.2023.34.e32. Epub 2022 Dec 15. PMID 36562136